CLINICAL TRIAL: NCT06392022
Title: The Effect of Having a Child Watch Musical Cartoons on Anxiety and Vital Signs During Rectal Irrigation
Brief Title: The Effect of Having a Child Watch Musical Cartoons
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: aysel kokcudogan (Other)
Responsible Party: Sponsor-Investigator, aysel kokcudogan, Assistant professor, Istanbul Medipol University Hospital
Organization: Istanbul Medipol University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: E-10840098-772.02-6325
Record Dates: First submitted 2024-04-20; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Child; Cartoon
Keywords: Anxiety; child; musical cartoons; vital signs
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Children in this group were shown musical cartoons during rectal irrigation.
  Interventions: Other: watching cartoons with music
- Control group (No Intervention): No additional intervention

INTERVENTIONS:
Other: watching cartoons with music — The purpose of this study was to evaluate the effect of watching musical cartoons on anxiety and vital signs in children undergoing rectal irrigation.
  Arms: Experimental group

SUMMARY:
The purpose of this study was to evaluate the effect of watching musical cartoons on anxiety and vital signs in children undergoing rectal irrigation. This study was a randomized controlled experimental trial. The study sample consisted of 40 children, 20 of whom were assigned to the experimental group and 20 to the control group. Data Collection Form, Vital Signs Evaluation Form, and Child Anxiety Scale-Stateness were used as data collection tools. Data collection tools were used in both groups before, during, and after the procedure. In addition, the experimental group was shown musical cartoons during the procedure.

DETAILED DESCRIPTION:
The present study was conducted as a randomized controlled experimental study to investigate the effect of watching musical cartoons on anxiety and vital signs in children undergoing rectal irrigation. Does watching musical cartoons during rectal irrigation have an effect on children anxiety and vital signs? The answer to the question has been sought.The study sample consisted of 40 children aged 4-10 years who met the inclusion criteria and whose parents provided written and verbal consent for their participation in the study after being informed at the Pediatric Surgery and Pediatric Urology Department of a public hospital affiliated to the Provincial Health Directorate of the Ministry of Health in Istanbul. Because of the high power requirement and the potential for loss to follow-up, the study was conducted with a total of 40 children, 20 assigned to the experimental group and 20 to the control group, who met the eligibility criteria and consented to participate. The children were randomly assigned to the control or experimental group. Children enrolled in the study were assigned to the experimental or control group using the https://www.calculatorsoup.com. Data Collection Form, Child Anxiety Scale-Stateness, and Vital Signs Evaluation Form were used as data collection tools.After obtaining institutional approval and written consent from parents after informing them and their children, data were collected by the investigators through a face-to-face interview that took approximately 11-20 minutes per child. The intervention to be applied to the experimental group was carried out by the investigator after informing the children and parents and obtaining their written consent.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 4-10 years
* Children who can count from one (1) to ten (10).
* Children who love cartoons with music.

Exclusion Criteria:

* Children without visual or hearing impairments
* Children without mental problems

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2021-12-13 (Actual); Primary Completion 2022-05-25 (Actual); Study Completion 2022-07-25 (Actual)

PRIMARY OUTCOMES:
Child Anxiety Scale-Stateness, | 10 minutes
  Child anxiety-state scale: Measures the anxiety state of children between the ages of 4-10.
  The level of anxiety increases as the scale rating progresses up to the top point.

SECONDARY OUTCOMES:
Vital signs evaluation | 10 minutes
  This form was developed by the investigators to record patients' vital signs (blood pressure, pulse rate, respiratory rate, body temperature) before, during, and after the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Aysel Kökcü Doğan, Study Director — Medipol University; Buse Tugcuoglu, Principal Investigator — Medipol University
Locations (1):
- Aysel Kokcu Dogan, Istanbul, Beykoz, Turkey (Türkiye)